CLINICAL TRIAL: NCT06006026
Title: The Safety of Ropivacaine Transversus Abdominis Plane Block Combined With Intravenous Lidocaine in Patients Undergoing Colorectal Cancer Surgery: a Single Center, Open Label Dose Escalation Study
Brief Title: The Safety of Ropivacaine TAP Block Combined With Intravenous Lidocaine in Patients Undergoing Colorectal Cancer Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Chunling Jiang, Professor, West China Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20201180HX
Record Dates: First submitted 2023-07-11; First posted 2023-08-23 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: Interventional Study Model: Sequential Assignment According to the principle of "the 3+3 design", 3 dose groups with 3 patients in each dose group will be set up. If no dose limited toxicity (DLT) is observed in three groups, a total of 9 patients will be included. If DLT is present in one dose group during dose escalation, 3 cases are amplified in this dose group; if no DLT is observed in 3 cases of amplification, proceed to the next dose group, and so on, up to 18 patients. DLT is defined as local anesthetic systemic toxicity. If blood samples cannot be obtained for any reasons, new patients will be recruited until there are at least 3 patients in each group with blood samples at every time point .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ropivacaine (Experimental): Patients will receive a TAP block using 1.5 mg/kg, 2.0 mg/kg or 2.5 mg/kg of ropivacaine. If there is no LAST (local anesthetic systemic toxicity) in the three subjects of 1.5 mg/kg group, the next three patients will receive 2.0 mg/kg of ropivacaine. Another three patients will receive 2.5 mg/kg of ropivacaine if there is no LAST in the three subjects of 2.0 mg/kg group. All subjects will be administered an i.v. bolus of lidocaine 2.0 mg/kg (given as an infusion for 10 min) after anaesthesia induction, then continuous infusion at 2 mg/kg/h until the end of surgery.
  Interventions: Drug: Ropivacaine Hydrochloride 10 MG/ML [Naropin]

INTERVENTIONS:
Drug: Ropivacaine Hydrochloride 10 MG/ML [Naropin] — According to the specified dosage, dilute 1% ropivacaine to 0.2% and inject 1/2 of the total amount on each side.

SUMMARY:
Many studies have confirmed the analgesic effect of intravenous infusion of lidocaine in abdominal surgery. Transversus abdominis plane (TAP) block is also often recommended for abdominal surgery. Ropivacaine TAP block and intravenous lidocaine infusion are important components of multimodal analgesia for colorectal surgery. However, both of them are the local anesthetics and the safety of combination is unknown, so investigators design the study to explore the safety of the synergistic application of ropivacaine TAP block and intravenous lidocaine infusion in patients undergoing colorectal surgery.

DETAILED DESCRIPTION:
Transversus abdominis plane (TAP) block is often recommended for abdominal surgery. Ropivacaine TAP block and intravenous lidocaine infusion are important components of multimodal analgesia for colorectal surgery. However, both of them are the local anesthetics and the safety of combination is unknown, so investigators design the study to explore the safety of the synergistic application of ropivacaine TAP block and intravenous lidocaine infusion in patients undergoing colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 65 years;
2. Patients who plan to undergo open/laparoscopic colorectal cancer resection surgery under general anesthesia;
3. American society of Anesthesiologists (ASA) physical status classification system I~II;

Exclusion Criteria:

1. Weight less than 40kg or more than 100kg;
2. Defects in the cardiac conduction system (II or III degree atrioventricular block) or cardiac dysfunction (LVEF<50%);
3. Severe liver dysfunction (ALT, AST, bilirubin 2.5 times higher than normal), renal dysfunction (creatinine clearance rate<60ml/min);
4. Allergies to experimental drugs;
5. Patients who are unable to communicate;
6. Participating in other clinical researchers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-08-28 (Actual); Primary Completion 2024-05-10 (Estimated); Study Completion 2024-05-20 (Estimated)

PRIMARY OUTCOMES:
The safety profile of combining ropivacaine and lidocaine | From administration of ropivacaine or lidocaine to postoperative 24 hours
  To observe signs of LAST, such as dizziness, light-headedness, metallic taste, peri-oral numbness, seizure activity or tinnitus, new-onset ECG irregularities, or intraoperative spike wave of EEG, et al.

SECONDARY OUTCOMES:
The plasma concentration of ropivacaine | From 10 min to 24h after the completion of bilateral TAP block
  Blood samples will be drawn at 10min, 20min, 30min, 45min, 60min, 90min, 2h, 4h, 6h, 12h and 24h after the completion of bilateral TAP block to measure the plasma ropivacaine concentration. All data will be tested for normality, then investigators will show the central tendency of the blood concentration of ropivacaine for all patients at each time point by means (standard deviation) or median (interquartile interval), the peak time and peak concentration of the blood concentration of ropivacaine. Investigators will also provide trends in the blood concentration of ropivacaine for each patient, and the concentration trend of blood drug concentration in each group of patients according to dose grouping.
The plasma concentration of lidocaine | From 10 min to 24h after the initiation of IV lidocaine.
  Blood samples will be drawn at 10min, 20min, 30min, 45min, 60min, 90min, 2h, 4h, 6h, 12h and 24h after the initiation of IV lidocaine to measure the plasma lidocaine concentration. All data will be tested for normality, then we will show the central tendency of the blood concentration of lidocaine for all patients at each time point by means (standard deviation) or median (interquartile interval), and the peak time and peak concentration of the blood concentration of lidocaine. Investigators will also provide trends in the blood concentration of lidocaine for each patient. and the concentration trend of blood drug concentration in each group of patients according to dose grouping.

CONTACTS AND LOCATIONS:
Overall Officials: Weiming Li, PhD, Principal Investigator — West China Hospital
Locations (1):
- West China hospital, Chengdu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou M, Yu F, Xu Y, Wu J, Luowu L, Tang Q, Hao X, Shao K, Ye M, Bo L, Zhou L, Jiang C. Combining ropivacaine transversus abdominis plane block with intravenous lidocaine infusion in adults undergoing colorectal cancer surgery: an open-label, dose-escalation exploratory trial. BMC Anesthesiol. 2025 Jul 22;25(1):357. doi: 10.1186/s12871-025-03225-5. PMID 40696274